CLINICAL TRIAL: NCT04637542
Title: The Effect of Mobile Learning on Student Success and Anxiety in Teaching the Genital System Anatomy
Brief Title: Anxiety Level of Nursing Students Before Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamiyet KIZIL (Other)
Responsible Party: Sponsor-Investigator, Hamiyet KIZIL, Lecturer Hamiyet KIZIL, University of Beykent
Organization: University of Beykent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1558
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Mobile Phone Use; Educational Problems; Anatomy
Keywords: gross anatomy education; high school education; mobile learning; anxiety level; genital system
MeSH Terms: conditions — Cell Phone Use

STUDY DESIGN:
Intervention Model Description: The research was designed in a randomized controlled experimental type. In the randomization of the study, using the Random.org website (Haahr, 2020) students were assigned to the experiment (mobile application group, n = 31) and control (traditional method group, n = 32) groups according to their numbers in the class list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Traditional) (Experimental): Application in the Control Group: After the theoretical lesson, the control group was taken to the Anatomy Laboratory. The laboratory consists of three application rooms, one control room and one analysis room. The "Anatomy of the Organs Forming the Genital System" was explained using an anatomical model of the genital system organs by a researcher responsible for the human anatomy course. Students were given time until the end of the lesson to work on the models. During this time, their questions were answered. At the end, all of the students were given a "State Inventory" by the researcher and asked to fill it in. Students were then asked to use textbooks and atlases to study for the "Knowledge Test (post-test)" which took place three days later.
  Interventions: Other: Mobile Learning
- Experimental Group (Mobile) (Experimental): Application in Experimental Group: After the theoretical lesson, students in the experimental group were taken to an empty classroom. The mobile application was installed on the smartphones of the students in the experimental group by the researchers and they were told not to share it with anyone until the end of the study. At the end of the study, the mobile application was also installed on the phones of the students in the control group due to ethical sensitivity. "Anatomy of Organs Forming the Genital System" was explained on the mobile application containing the genital system organs. The students were allowed to ask questions and the questions were answered. Afterwards, all students in the experimental group were given a "State Inventory" by the researcher and asked to fill it in. Students were then asked to study using the "genitalsystem.apk" mobile application until the "Knowledge Test (post-test)" which took place three days later.
  Interventions: Other: Mobile Learning

INTERVENTIONS:
Other: Mobile Learning — The necessary interviews and correspondences were carried out in order to conduct the research. Permission was obtained from Health Sciences University Istanbul Training and Research Hospital Clinical Research Ethics Committee. The purpose of the study was explained to the students as per the sample criteria and their consents were obtained. All of the students participating in the study attended four hours of theoretical lessons in the classroom related to anatomy of the genital system. Following the theoretical training, students were divided into experiment (mobile application) and control (genital organ model) groups. Both groups where then given the "Structured Student Presentation Form", "Status and trait anxiety inventory" and "Knowledge Examination (pre-test)" on paper.
  The didactic content prepared for the institution's standard curriculum (control group) or mobile learning is similar for both training methods.

SUMMARY:
The widespread use of smartphones today has led to the emergence of new ways of teaching, such as mobile learning. This research was conducted to determine the effectiveness of mobile learning on students' success and anxiety in teaching the anatomy of the genital system.

This research is a randomized controlled experimental study conducted with students who took anatomy classes at a private university between November-December 2018.The sampling consisted of 63 students who met the sampling criteria of the study and who were given permission to participate in the research after the information was explained. Control (n=31) and experimental group (n = 32) were determined by randomization using simple numbers table. The mobile application developed for the experimental group was installed on the students' android devices with the extension "genitalsystem.apk".The anatomy of the genital system was taught to the control group with a standard curriculum and to the experimental group via the mobile learning.

In this context, the study hypothesizes that mobile learning is effective in teaching the anatomy of the genital system, and that the success levels of students who receive an education through mobile learning are higher and their anxiety levels are lower than those who receive education through traditional methods.

DETAILED DESCRIPTION:
This research was conducted to determine the effectiveness of mobile learning on students' success and anxiety in teaching the anatomy of the genital system.

Participants The research is a randomized controlled experimental study. This study was conducted with students who took anatomy lessons at a private university between November and December 2018. Power analysis to determine the number of students to form the research sample was performed using NCSS-PASS statistical package (NCSS, LLC., Kaysville, UT). In order to make a study with this analysis P ≤ 0.1 levels, the number of samples was decided to be 60. As a result, the sample of the research; By explaining the purpose of the study, a total of 63 students who was allowed to participate in the post-informative research and meet the sample criteria of the research was formed. Sampling criteria; the student is not (1) not a graduate of a health vocational high school, (2) has not previously been trained in mobile learning, (3) has taken the anatomy course for the first time, (4) received written and verbal permission for participation in the study.

Designed of Study and Randomization The research was designed in a randomized controlled experimental type. In the randomization of the study, using the Random.org website, students were assigned to the experiment (mobile application group, n = 31) and control (traditional method group, n=32) groups according to their numbers in the class list.

Data Collection Tools The research data were collected with "Structured Student Information Form", "State and Trait Anxiety Inventory", "Knowledge Examination on the anatomical structure of the genital system".

Structured Student Introduction Form The socio-demographic characteristics of the student identification form, such as the students' age, gender as well as data on educational status are included. It consists of five questions in total.

State and Trait Anxiety Inventory In the research, two different scales were applied to the students. These are the State Anxiety Scale (STAI FORM TX - I) and the Trait Anxiety Scale (STAI FORM TX - 2). The scale was developed in 1970 by Speilberger et al. The adaptation and adjustment of the scales into Turkish was done by Necla Öner and Ayhan LeCompte in 1983. It consists of 20 items in both scales and is graded in a four-point Likert style. Scoring is done between 1-4. The answer options collected in four classes in the state anxiety scale (WHO), (1) None, (2) A little, (3) A lot, and (4) Completely. In the Trait Anxiety Scale (SAD) options (1) Almost never, (2) Sometimes, it is (3) Much time and (4) Almost always. The scores obtained from both scales theoretically range from 20 to 80. Larger scores mean high anxiety levels while, smaller score means low anxiety level. In this study, Cronbach's alpha value of the scale was found to be 0.95.

Knowledge examination on the anatomical structure of the genital system:

The genital system examination prepared according to the literature consists of 22 questions including the anatomical structure. The knowledge examination contains the names of the anatomical structures of the genital system on the figure. It was created by taking color copies of the images on paper. The lowest score that can be obtained from the knowledge examination is determined as "0" and the highest score as "100".

Different learning methods were used in both groups, but the examination was conducted in the same format. The pre-test and post-test examinations contain the same questions. An equal number of questions were asked about male and female genital system issues.

Collection of Data The necessary interviews and correspondences were carried out in order to conduct the research. Permission was obtained from Health Sciences University Istanbul Training and Research Hospital Clinical Research Ethics Committee. The purpose of the study was explained to the students as per the sample criteria and their consents were obtained. All of the students participating in the study attended four hours of theoretical lessons in the classroom related to anatomy of the genital system. Following the theoretical training, students were divided into experiment (mobile application) and control (genital organ model) groups. Both groups where then given the "Structured Student Presentation Form", "Status and trait anxiety inventory" and "Knowledge Examination (pre-test)" on paper.

The didactic content prepared for the institution's standard curriculum (control group) or mobile learning is similar for both training methods.

Application in the Control Group: After the theoretical lesson, the control group was taken to the Anatomy Laboratory. The laboratory consists of three application rooms, one control room and one analysis room. The "Anatomy of the Organs Forming the Genital System" was explained using an anatomical model of the genital system organs by a researcher responsible for the human anatomy course. Students were given time until the end of the lesson to work on the models. During this time, their questions were answered. At the end, all of the students were given a "State Inventory" by the researcher and asked to fill it in. Students were then asked to use textbooks and atlases to study for the "Knowledge Test (post-test)" which took place three days later.

Application in Experimental Group: After the theoretical lesson, students in the experimental group were taken to an empty classroom. The mobile application was installed on the smartphones of the students in the experimental group by the researchers and they were told not to share it with anyone until the end of the study. At the end of the study, the mobile application was also installed on the phones of the students in the control group due to ethical sensitivity. "Anatomy of Organs Forming the Genital System" was explained on the mobile application containing the genital system organs. The students were allowed to ask questions and the questions were answered. Afterwards, all students in the experimental group were given a "State Inventory" by the researcher and asked to fill it in. Students were then asked to study using the "genitalsystem.apk" mobile application until the "Knowledge Test (post-test)" which took place three days later

Mobile Application Development Stage The use of technology in education helps students with their individual learning development. However, for a successful integration of technology into education, multiple design principles should be considered. In this context, the "Mayer Multimedia Design Principles" were considered in designing the mobile application developed within the scope of the research.

The mobile application was developed with Adobe Flash CS6 for Android devices with the extension "genitalsystem.apk". The application was uploaded to the smartphones of the experimental group by the researcher.

The homepage of the mobile application consists of five sections: the male genital system, the female genital system, the path followed by the sperm, the path followed by the ovum and the purpose of the mobile application.

The male genital system is divided into two sections, presented on the application as two separate pages: internal genital organs and external genital organs. Both pages on the mobile application are operated in the same way: the user presses on the red dots that are programmed on the page, which makes the anatomical names of the organs appear on a rectangular area at the top of the screen.

The female genital system is divided into two sections, presented on the application as two separate pages: internal genital organs and external genital organs. Both pages on the mobile application are operated in the same way: the user presses on the red dots that are programmed on the page, which makes the anatomical names of the organs appear on a rectangular area at the top of the screen.

The page on the mobile application detailing the path followed by the sperm features an animation that shows the section from the production of sperm to the woman's external genital area. The users can start, stop or watch the animation whenever they want. During the animation of the path followed by the sperm, the name of the anatomical region the sperm has reached appears at the top of the screen.

The page on the mobile application detailing the path followed by the ovum features an animation that shows the section from the production of ovum to zygote formation. The users can start, stop or watch the animation whenever they want. During the animation of the path followed by the ovum, the name of the anatomical region the ovum has reached appears at the top of the screen.

On the purpose of the mobile application page, users can access the sources of the information provided by researches for the purposes of mobile use and the information used for the mobile application.

Statistical Methods A licensed SPSS statistical package, version 25.0 for Windows (IBM Corp) was used for data analysis. The distribution of the demographic information of the participants by groups was analyzed by chi-square analysis. Whether the average age varies significantly between the groups was investigated with the t-test in independent groups. Normal distribution among the groups in the state anxiety and trait anxiety inventory was analyzed with the Kolmogrov Smirnov and Shapiro Wilks test and it was observed that they were compatible with the normal distribution. Pretest-posttest comparisons were examined with t-test in dependent groups and comparison of measurements by study groups with t-test in independent groups. Regardless of whether the state and trait anxiety levels had a significant effect on the knowledge score, regression analysis was examined. Results were evaluated at 95% confidence interval and significance level at P < 0.05.

Ethical and Legal Aspects of the Research The necessary interviews and correspondences were carried out in order to conduct the research. Approvals were obtained from the institution and ethics committee (S.U.U Istanbul Training and Research Hospital Clinical Research Ethics Committee- No: 1558 /07.12.2018). The students who formed the research sample have been informed about the purpose, plan, duration and procedures to be done. Therefore, informed consent has been obtained for their participation in the research through their own willingness and on the principle of volunteering.

ELIGIBILITY:
Inclusion Criteria:

* the student is not a graduate of a health vocational high school,
* the student has not previously been trained in mobile learning,
* the student has taken the anatomy course for the first time,
* the student received written and verbal permission for participation in the study.

Exclusion Criteria:

* the student is a graduate of a health vocational high school,
* the student has previously been trained in mobile learning, ,
* the student has taken the anatomy course for the second time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Success level | 2 Months
  The student were informed abaout Knowledge examination on the anatomical structure of the genital system

SECONDARY OUTCOMES:
anxiety level | 2 Months
  The student were informed abaout State and Trait Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, RN Msc, Principal Investigator — Beykent University
Locations (1):
- Hamiyet Kızıl, Istanbul, Beykent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward PJ, Walker JJ. The influence of study methods and knowledge processing on academic success and long-term recall of anatomy learning by first-year veterinary students. Anat Sci Educ. 2008 Mar-Apr;1(2):68-74. doi: 10.1002/ase.12. PMID 19177384
- [Background] Waterston SW, Stewart IJ. Survey of clinicians' attitudes to the anatomical teaching and knowledge of medical students. Clin Anat. 2005 Jul;18(5):380-4. doi: 10.1002/ca.20101. PMID 15971223
- [Background] Wallace S, Clark M, White J. 'It's on my iPhone': attitudes to the use of mobile computing devices in medical education, a mixed-methods study. BMJ Open. 2012 Aug 24;2(4):e001099. doi: 10.1136/bmjopen-2012-001099. Print 2012. PMID 22923627